CLINICAL TRIAL: NCT05441150
Title: Effect of Intraoperative Intravenous Ketamine Infusion on Postoperative Analgesia in Right Hepatectomy of Living Liver Donors
Brief Title: Intravenous Ketamine Infusion on Postoperative Analgesia of Living Liver Donors
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Mehmet Ali Erdoğan, Inonu University, School of Medicine, Department of Anaesthesiology and ReanimationMalatya, Turkey, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ketamin-Postopanalgesia
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Liver Failure; Liver Transplant; Complications; Post Operative Pain
Keywords: Living liver donor; Liver; Transplantation; postoperative pain; ketamine
MeSH Terms: conditions — Liver Failure; Pain, Postoperative | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Group (Active Comparator): Patients who received low-dose ketamine infusion
  Interventions: Drug: Low dose ketamine infusion
- Control group (Sham Comparator): Patients who received 0.9% Sodium Chloride Solution, Intravenous, (NaCl) infusion
  Interventions: Drug: 0.9% NaCl infusion

INTERVENTIONS:
Drug: Low dose ketamine infusion — Administering low-dose ketamine infusion to the patient under general anesthesia for Ketamine Group.
  Other Names: Ketamine
  Arms: Ketamine Group
Drug: 0.9% NaCl infusion — Same dose of 0.9% NaCl infusion as the dose of ketamine for Control Group.
  Other Names: Saline
  Arms: Control group

SUMMARY:
Because of the insufficiency of cadaveric organs and increasing need for organs, the interest in living donor liver transplantation have been greatly increased. The relative reduction of the remaining liver after the operation in Living Liver Donors makes it difficult and compelling to choose a very effective and very safe method in the management of postoperative analgesia.

Opioids are the main agents used in the postoperative analgesia of Live Liver Donors. Opioids have serious side effects such as respiratory depression, apnea, circulatory collapse, coma, and death. Both short-term and long-term administration of opioids cause acute opioid-induced hyperalgesia.

Ketamine, an NMDA receptor antagonist, has been hypothesized to counter opioid tolerance and NMDA receptor-mediated central sensitization. Various studies and systematic reviews have shown that low-dose ketamine has an opioid-sparing effect in all surgical patients.

Although low-dose ketamine has been shown to be beneficial overall in relieving pain, it is unclear whether it has an identified benefit in hepatectomy cases. The aim of this clinical trial was to evaluate the effect of low-dose ketamine administration on postoperative analgesia in living donor liver donors undergoing right hepatectomy procedure.

DETAILED DESCRIPTION:
Liver transplantation is the only treatment for end-stage liver failure. The insufficiency of cadaveric organs and the inability to meet the increasing need for organs with cadaveric transplantations have greatly increased the interest in living donor liver transplantation. The relative reduction of the remaining liver after the operation in Living Liver Donors makes it difficult and compelling to choose a very effective and very safe method in the management of postoperative analgesia.

Opioids are the main agents used in the postoperative analgesia of Live Liver Donors. Opioids have serious side effects such as respiratory depression, apnea, circulatory collapse, coma, and death. Both short-term and long-term administration of opioids cause acute opioid-induced hyperalgesia.

There is evidence that opioid tolerance can occur in the dorsal root ganglion through N-methyl-D-aspartate (NMDA) receptor activation. Ketamine, an NMDA receptor antagonist, has been hypothesized to counter opioid tolerance and NMDA receptor-mediated central sensitization. Low-dose ketamine is an effective adjuvant in painful orthopedic procedures that reduces pain and opioid need, especially in the first 24 hours after the procedure. Various studies and systematic reviews have shown that low-dose ketamine has an opioid-sparing effect in all surgical patients.

Although low-dose ketamine has been shown to be beneficial overall in relieving pain, it is unclear whether it has an identified benefit in hepatectomy cases. The aim of this randomized placebo-controlled clinical trial was to evaluate the effect of low-dose ketamine administration on postoperative analgesia in living donor liver donors undergoing a painful right hepatectomy procedure.

ELIGIBILITY:
Inclusion Criteria:

* living liver donors, aged 16-65 years, who are scheduled for right hepatectomy will be included in the study.

Exclusion Criteria:

* to use opioid medications before surgery,
* trauma,
* body mass index (BMI) >35,
* unstable ischemic heart disease,
* increased intracranial or intraocular pressure,
* lactation,
* to have an allergic to ketamine, morphine, propofol or remifentanil,
* psychiatric illness, patient-controlled analgesia (PCA)
* unwillingness or inability to use the device
* inability to use the numerical rating scale (NRS).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 24 hour
  To determine the cumulative opioid consumption at the end of 24 hours in patients who received low-dose ketamine or 0.9% NaCl infusion.

SECONDARY OUTCOMES:
Postop Sedation Score | Postoperative 1 hour
  Postop Sedation Score (0-3): sedation was measured on a scale of 0 to 3 0: fully awake; 1: lightly sedated, rarely sleepy and easily aroused; 2: moderately sedated, often sleepy and easily aroused; 3; severely sedated, sleepy and difficult to wake up
postoperative complications | 24 hour
  postoperative complications: pruritus, vomiting, hallucination

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu university, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I am hesitant to share the data before completing the study. However after end of the study I might consider sharing